CLINICAL TRIAL: NCT03809975
Title: Collaborative Model of Care Between Orthopaedics and Allied Healthcare Professionals Trial (CONnACT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: University of Southern Denmark (Other); Nanyang Technological University (Other); Singapore General Hospital (Other); University of Sydney (Other)
Responsible Party: Principal Investigator, Bryan Tan, Senior Resident, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTF_JUL2017_I_C2_CQR_01; 2018/00408 (Other: NHG RDO - DSRB)
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthritis
Keywords: Knee; Osteoarthritis; Model of care; Multi-disciplinary
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Current model of care
  Patients will undergo the current standard of care in the Orthopaedic Outpatient Clinic in Tan Tock Seng Hospital. Patients will undergo routine consultation with an orthopaedic surgeon and will be provided with standard treatment as necessitated based on the assessment of the orthopaedic surgeon. Subsequent follow up appointments will be scheduled at the discretion of the orthopaedic surgeon. Patients will be referred to the physiotherapists, dietitian and psychologists as necessary for regular or adhoc sessions at the discretion of the allied health professional.
  Interventions: Other: Current model of care
- Intervention Arm (Experimental): Multidisciplinary Community Program
  Community based, personalized, structured, 12-week multidisciplinary program that includes Orthopaedics, Physiotherapy, Dietitics, Psychology interventions. This intervention involves the use of formal assessment such as BMI and psychological questionnaires to determine the need for dietetics or psychological intervention. In addition, there are educational sessions to improve patient's understanding of osteoarthritis and improve their activation level. An optional support group session will be arranged at approx. 3-4 months after completion of the 12-week intervention program to improve sustainability of treatment effect.
  Interventions: Other: Multidisciplinary Community Program

INTERVENTIONS:
Other: Multidisciplinary Community Program — Patient will undergoes 12 weeks of structured and personalized multidisciplinary community-based program, which consists of Physiotherapy, Dietetics and Psychology sessions. Patients will also attend 2 educational sessions. Physiotherapy and educational sessions are mandatory for all participants, while the need for dietetics and psychological interventions are determine using individual's BMI measurements and psychological questionnaires.
  Inclusion criteria:
  Dietetics: 23.5 < BMI <32.5; Psychology: PEG > 4 or PHQ-4 > 5 or PAM level < 3
  Arms: Intervention Arm
Other: Current model of care — No controlled set of treatment assigned to patient. It is based totally on the discretion of the attending clinicians. It will generally contain an unspecific number of physiotherapy sessions. Other allied health involvement such as dietetics and psychological interventions will be on an ad hoc basis. In some cases, the orthopaedic surgeon may recommend for surgery.
  Arms: Control Arm

SUMMARY:
Osteoarthritis knee is the leading cause of chronic disability among older adults. Our current model of care is doctor-centric and inefficient leading to suboptimal use of allied health intervention for effective lifestyle and behaviour changes resulting in potentially, unnecessary surgery.

The study is designed using an effectiveness-implementation hybrid study design utilizing a mixed methods approach. The hybrid study has dual aims. The primary aim is to evaluate the clinical effectiveness (pain, function and quality of life) of a 12-week multidisciplinary (Orthopaedics, Physiotherapy, Dietetics, Psychology) personalized, community-based program for patients with knee osteoarthritis through a randomized-controlled trial. The secondary aim is to obtain data that will inform the context for implementation and guide future wider scale application. The investigators hypothesize that this multidisciplinary program is clinically more effective in the treatment of knee osteoarthritis at 12 months compared to standard care.

DETAILED DESCRIPTION:
BACKGROUND With a rapidly aging population, osteoarthritis is expected to become the 4th leading cause of global disability by 2020. Established guidelines for knee osteoarthritis strongly advocate lifestyle changes, such with exercises and weight loss as first line of treatment, whilst reserving surgery as the last resort. Our current model of care is doctor-centric and inefficient leading to suboptimal use of allied health intervention for effective lifestyle and behaviour changes resulting in potentially, unnecessary surgery. Redesigning the model of care by moving away from costly surgical treatment through the optimization and synergizing of proven non-surgical treatments is key to deliver value-based care.

AIMS AND HYPOTHESIS Primary Aim and Hypothesis. Evaluate the clinical effectiveness (pain, function and quality of life) at 12 months of a personalized, community based 3-month multidisciplinary program (Orthopaedics, Physiotherapist, Dietitian and Psychologist) as compared with usual care for patients with knee osteoarthritis. The investigators hypothesize that patients with knee osteoarthritis who undergo a personalized, community based 3-month multidisciplinary program will have better pain, function and quality of life scores at 12 months post initiation of program compared to patients who undergo usual care.

Secondary Aim. Evaluate the cost effectiveness of a personalized, community based 3-month multidisciplinary program (Orthopaedic, Physiotherapist, Dietitian and Psychologist) for patients with knee osteoarthritis. Qualitative assessment of the acceptability, feasibility and scalability of such a program

METHODOLOGY The study will be conducted as a single centre, single-blinded, gender stratified, block permutated randomized controlled trial using a mixed method approach (quantitative and qualitative), comparing a proposed new multidisciplinary personalized community-based model of care and the current model of care.

Patients with suspected knee osteoarthritis who are referred from the Polyclinics in the primary healthcare setting to the Tan Tock Seng Hospital Orthopaedic Specialist Outpatient Clinic. Patients will then be evaluated based on the inclusion and exclusion criteria and subsequently invited to join the study if eligible. Consent for participation into the study will be obtained prior to randomization. Randomization will be done via gender stratified permutated block randomization.

ECONOMIC EVALUATION An economic evaluation from a societal perspective will be undertaken to determine the cost effectiveness of the intervention. The incremental cost effectiveness ratio of this multidisciplinary non-surgical community-based program for knee osteoarthritis compared to routine care will be determined. Cost data will be collected via questionnaires and hospital databases to estimate both the direct medical, direct non-medical and indirect cost. Indirect cost of health-related productivity loss due to knee osteoarthritis will be calculated using a human capital approach. The primary measure of health benefit will be Quality of Life Years measure using the EQ-5D.

QUALITATIVE COMPONENT The qualitative component of our study will employ several qualitative methods such as focus group discussions and individual interviews with a variety of subjects including both patients and stakeholders. The focus will on identifying the potential barriers and facilitators to implementing and upscaling the intervention.

ELIGIBILITY:
Inclusion Criteria

1. National Institute for Health and Care Excellence (NICE) clinical criteria for knee osteoarthritis
2. Radiographic severity of knee osteoarthritis - Kellgren Lawrence Score > 1
3. Knee Injury and Osteoarthritis Outcome Score (KOOS4) ≤ 75
4. Independent community ambulator with or without walking aid
5. Age ≥ 45 years old
6. Conversant in English/Chinese
7. Subject will need to fulfill all the inclusion criteria for eligibility.

Exclusion Criteria

1. Alternative diagnosis to knee osteoarthritis e.g. referred pain from the spine or hip
2. Secondary arthritis e.g. inflammatory, post-traumatic
3. Inability to comply with study protocol e.g. cognitive impairment
4. Previous knee arthroplasty on the symptomatic knee
5. Wheelchair bound patients
6. Any other medical condition that study team determines may interfere with study involvement

Ages: 45 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcomes Score (KOOS4) | Assessed at baseline, 3 months, 6 months, 12 months
  Change in disease specific pain and functional outcome scores between patients undergoing the multidisciplinary community program and the current model of care will be evaluated. A composite score of the following subscales will be calculated using the averaged score - Pain, Symptoms, Activities of Daily Living and Quality of Life will be calculated. Scores between 0 and 100 represent the percentage of total possible score achieved, with zero representing extreme knee problems and 100 representing no knee problems.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcomes Score (KOOS) subscales - Pain, Symptoms, Activities of Daily Living, Sports/Recreational Activities, Quality of Life | Assessed at baseline, 3 months, 6 months, 12 months
  The five patient-relevant subscales of KOOS are scored separately: KOOS Pain (9 items); KOOS Symptoms (7 items); KOOS ADL (17 items); KOOS Sport/Rec (5 items); KOOS QOL (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems
EuroQol-5 Dimensions (EQ-5D) | Assessed at baseline, 3 months, 6 months, 12 months
  EuroQol-5 Dimensions (EQ-5D) which consist of 2 dimensions, the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS will be used as a quantitative measure of health outcome.
Functional Assessment - 30s chair stand test | Assessed at baseline, 3 months, 6 months, 12 months
  To test leg strength and endurance. Total number of repetitions completed in 30 seconds is recorded.
Functional Assessment - 40m fast-paced walk test | Assessed at baseline, 3 months, 6 months, 12 months
  Measure of patient's walking speed. Time taken to complete 40 meters walk will be recorded in seconds.
Functional Assessment - 4 stairs climb test | Assessed at baseline, 3 months, 6 months, 12 months
  To assess the strength, balance and agility through ascending and descending a set number of steps. Time to ascend and descend steps (excluding turning around time) is recorded separately in seconds. Overall time taken (including the turn around time) to ascend and descend stairs is also recorded.
Functional Assessment - Timed up and go test | Assessed at baseline, 3 months, 6 months, 12 months
  To assess patient's mobility and balance through the patient's ability to rise from a seated position to walk around a cone 3 meters away and return to the seated position. Time taken to perform the test in fast walking pace will be recorded in seconds.
Patient Health Questionnaire 4 (PHQ-4) | Assessed at baseline, 3 months, 6 months, 12 months
  Measurement for depression and anxiety rated on a 4 point Likert-type scale. 0 refers to 'Not at all'; 3 refers 'Nearly everyday'. Total score is determined by adding together the scores of each of the 4 items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12).
  Total score ≥3 for first 2 questions suggests anxiety. Total score ≥3 for last 2 questions suggests depression.
Patient Activation Measure (PAM) | Assessed at baseline, 3 months, 6 months, 12 months
  Measures patients on a 0-100 scale and can segment patients into one of four activation levels along an empirically derived continuum. Each activation level reveals insight into an array of health-related characteristics, including attitudes, motivators, behaviors, and outcomes.
Pain, Enjoyment, General Activity Scale (PEG) | Assessed at baseline, 3 months, 6 months, 12 months
  Measures the pain intensity and interference level using a three-item scale. Scale of 0 to 10 is used for each item. 0 refers 'no pain'; 10 refers 'worse pain'. Add the responses to the three questions, then divide by three to get a mean score (out of 10) on overall impact of points.
Body Mass Index (BMI) | Assessed at baseline, 3 months, 6 months, 12 months
  Assessed if patient achieved weight loss during the study period. Weight and height of patient will be measured in m and kg respectively. Weight and height will be combined to report BMI in kg/m^2
Total Knee Replacement | Assessed at 3 months, 6 months, 12 months
  Indicates if the patient undergoes a total knee replacement at any time during the study period.

OTHER OUTCOMES:
Cumulative Analgesia Consumption Score (CACS) | Assessed at baseline, 3 months, 6 months, 12 months
  Objective measurement of patient's analgesics average weekly consumption based on the quantity multiplied by the category of analgesic medication according to the WHO pain relief ladder(1 point - non-opioid, 2 points - mild opioid, 3 points - strong opioid) in order to calculate a total score.
Semi-Quantitative Food Frequency Questionnaire (FFQ) | Assessed at baseline, 3 months, 6 months, 12 months
  Understand the eating habits and dietary choice over time. 64 question questionnaire looking at the frequency of food consumption in different food group on a 5 point scale ranging from less than 3 times a month to more than once a day.
Sports Injury Rehabilitation Adherence Scale (SIRAS) | Assessed after each physiotherapist session
  A measurement of the patient's compliance level to exercises done by the attending therapist. 3 question questionnaire with an answering scale of 1 to 5. Total score is derived from adding the 3 scores up.
Global perceived effect (GPE) | Assessed at 3 months, 6 months, 12 months
  Patient will be asked to rate their overall recovery on a 7-point Likert scale. 1 refers to 'Very much improved'; 7 refers to 'Very much deteriorated'.
Patient Acceptable Symptom State (PASS) | Assessed at 3 months, 6 months, 12 months
  A single-question used to assess patient's satisfaction in the treatment. Response will be either yes or no."When you think of your knee function, will you consider your current condition as satisfying? By knee function, you should take into account your activities of daily living, sport and recreational activities, your pain and other symptoms and your quality of life"
Patient-reported Treatment failure | Assessed at 3 months, 6 months, 12 months
  Patient who answers 'no' to PASS will be ask to determine if they consider the treatment to have failed. Response will be 'yes' or 'no'. "Would you consider your current state as being so unsatisfactory that you consider the treatment to have failed?"
Costs | Assessed at 3 months, 6 months, 12 months
  Cost questionnaire measuring the direct and indirect costs
Adverse Events | Assessed at 3 months, 6 months,12 months
  Adverse events (AE) and serious adverse events (SAE) will be recorded at all follow-ups by asking the participants about potential AEs using open-probe questioning to ensure that all AEs are recorded. AEs will be categorized into index knee or other sites and will be recorded and assessed for severity independent of whether or not there is a causal relationship with study treatments.
University of California, Los Angeles(UCLA) activity score | Assessed at baseline, 3 months, 6 months and 12 months
  1 question survey to understands patient physical activity level from a scale of 1(wholly inactive) to 10(regular participation in impact sports).

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Tan, MBBS, MRCS, Principal Investigator — Tan Tock Seng Hospital; Soren Skou, PT, PhD, Study Chair — University of Southern Denmark; Josip Car, MD, PhD, Study Chair — Nanyang Technological University; Julian Thumboo, MBBS, FRCP, Study Chair — Singapore General Hospital; David Hunter, MBBS, PhD, Study Chair — University of Sydney
Locations (2):
- Singapore (2):
  - St Luke Eldercare (AMK), Singapore
  - Tan Tock Seng Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tan BY, Yang SY, Pereira MJ, Tan CY, Lim CJ, Ng JP, Lee KT, Pua YH, Briggs AM, Hunter DJ, Skou ST, Thumboo J, Car J. Collaborative model of care between orthopaedics and allied healthcare professionals (CONNACT) in knee osteoarthritis: Effectiveness-implementation hybrid randomized controlled trial of a community-based, multidisciplinary, stratified intervention. Osteoarthritis Cartilage. 2024 Aug;32(8):972-981. doi: 10.1016/j.joca.2024.04.018. Epub 2024 May 6. PMID 38710437
- [Derived] Tan BY, Pereira MJ, Yang SY, Hunter DJ, Skou ST, Thumboo J, Car J. Collaborative model of care between Orthopaedics and allied healthcare professionals in knee osteoarthritis (CONNACT): study protocol for an effectiveness-implementation hybrid randomized control trial. BMC Musculoskelet Disord. 2020 Oct 16;21(1):684. doi: 10.1186/s12891-020-03695-3. PMID 33066746
- [Derived] Tan BY, Ding BTK, Pereira MJ, Skou ST, Thumboo J, Car J. Collaborative model of care between Orthopaedics and allied healthcare professionals trial (CONNACT) - a feasibility study in patients with knee osteoarthritis using a mixed method approach. BMC Musculoskelet Disord. 2020 Sep 4;21(1):592. doi: 10.1186/s12891-020-03611-9. PMID 32887594